CLINICAL TRIAL: NCT07250191
Title: The Acute Effects of Energy and Carbohydrate Restriction on Postprandial Metabolism
Brief Title: The Effects of 24-hour Fasting or Carbohydrate Restriction on Postprandial Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Guoda Karoblyte, Doctoral Researcher, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0590
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Glucose and Lipid Metabolism
Keywords: carbohydrate restriction; fasting; intermittent energy restriction
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse; Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Habital control diet (No Intervention): 100% of energy requirements, ≥150 carbohydrate/day
- Fasting (Experimental): No energy intake
  Interventions: Behavioral: Fasting
- Carbohydrate Restriction (Experimental): 100% of energy requirements, ≤20g carbohydrate
  Interventions: Behavioral: Carbohydrate restriction

INTERVENTIONS:
Behavioral: Fasting — No food intake for 24 hours
  Arms: Fasting
Behavioral: Carbohydrate restriction — Restriction of dietary carbohydrate to ≤5% of total energy intake for 24 hours
  Other Names: Ketogenic diet
  Arms: Carbohydrate Restriction

SUMMARY:
Most individuals spend the majority of the day in a fed state, making postprandial blood glucose and lipid regulation a central component of metabolic health. Short periods of fasting or reduced carbohydrate intake can occur frequently in daily life, whether through intentional dietary practices (e.g. intermittent fasting), cultural or religious traditions, or unstructured eating patterns. These periods can induce measurable metabolic changes, but the acute effects of a single 24-hour period of fasting or carbohydrate restriction on postprandial metabolism upon refeeding remain poorly characterised.

This study will examine how 24 hours of either complete fasting or low carbohydrate intake without energy restriction influence postprandial blood glucose and lipid concentrations, as well as related metabolic markers, in healthy adults, in comparison to a habitual high carbohydrate control diet. Participants will complete all three conditions in a randomised order, consuming a standardised meal test after each 24-hour condition. Repeated blood sampling and gas exchange measurements will be carried out to assess postprandial metabolic responses.

The aim of this study is to characterise whether acute periods of fasting and low carbohydrate restriction elicit distinct or comparable alterations in postprandial metabolic responses. A clearer understanding of these acute physiological effects can help inform how variations in eating patterns influence glucose and lipid handling in individuals without metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-40 years
* Have a BMI of 18.5-29.9 kg/m2

Exclusion Criteria:

1. Diagnosed with any major chronic conditions (e.g. type 2 diabetes, coronary heart disease, cancer, chronic kidney disease, etc.)
2. Use of medication that may interfere with study outcomes (e.g. glucose or lipid-lowering medications)
3. Currently or recently pregnant (within last 6 months), planning to get pregnant or currently lactating
4. Has a habitually low carbohydrate intake (<150g carbohydrates/day)
5. Current or previous eating disorder
6. Has donated more than 500ml of blood in the last 3 months prior to the initial laboratory visit
7. Insufficient mental capacity or language skills to independently understand and follow the study protocol
8. Has an irregular sleeping pattern (e.g. due to undertaking night-shift work)
9. Any other condition, concurrent intervention or behaviour deemed either to pose undue personal risk to the participant or to introduce bias into the experiment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Triglyceride Concentration | After each 24-hour dietary condition
  Plasma triglyceride concentrations assessed at baseline and postprandially for 2 hours after a mixed meal test
Glucose Concentration | After each 24-hour dietary condition
  Plasma glucose concentrations assessed at baseline and postprandially for 2 hours after a mixed meal test

SECONDARY OUTCOMES:
Insulin Concentration | After each 24-hour dietary condition
  Plasma insulin concentrations assessed postprandially for 2 hours after a mixed meal test
Non-esterified Fatty Acid Concentration | After each 24-hour dietary condition
  Plasma non-esterified fatty acid concentrations assessed at baseline and postprandially for 2 hours after a mixed meal test
Beta-hydroxybutyrate Concentration | After each 24-hour dietary condition
  Plasma beta-hydroxybutyrate concentrations assessed at baseline and postprandially for 2 hours after a mixed meal test
Substrate Oxidation | After each 24-hour dietary condition
  Lipid and carbohydrate oxidation assessed via indirect calorimetry at baseline and during 2-hour mixed meal test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No